CLINICAL TRIAL: NCT04278521
Title: Mechanism of Action of Transcranial Magnetic Stimulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joan A Camprodon, MD MPH PhD, Chief of Division of Neuropsychiatry, Director of TMS Clinic, Director of Lab for Neuropsychiatry and Neuromodulation, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P001835
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder; Depression
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Unipolar Depression (Other): Patients diagnosed with unipolar depression.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial magnetic stimulation uses a rapidly changing magnetic field to induce current in brain tissue non-invasively. It is common procedure in both clinical and research settings, and it has well established guidelines for safe an ethical use which maximize safety for all subjects.
  Other Names: TMS

SUMMARY:
This is an observational neuroimaging study assessing the effects of TMS on the brains of patients with unipolar depression.

DETAILED DESCRIPTION:
This project aims to use functional connectivity magnetic resonance imaging (fcMRI) to study patients with unipolar depression receiving TMS. Patients will be scanned before and after a full course of TMS and clinical measures for depression severity and memory will be obtained at the same times.The project has the following aims and hypothesis: (1) to determine the therapeutic antidepressant mechanism of action of TMS at the circuit level (2) to study the use of fcMRI as a state biomarker for depression (3) to study the use of fcMRI as a predictor of response for depression.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 18-80
2. DSM-IV diagnosis of Depressive Episode
3. Patients requiring TMS treatment as part of their psychiatric care

Exclusion Criteria:

1. Comorbid DSM-IV primary diagnoses of schizoaffective disorder, schizophrenia or dementia.
2. Substance use disorder (abuse or dependence) with active use within the last 3 months
3. Severe or unstable medical illness.
4. MRI contraindications as determined by MGH department of radiology.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in Functional Connectivity of Key Nodes in Depression | Through Treatment Completion, Average of 6 Weeks
  Measured by Magnetic Resonance Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Joan Camprodon, MD, PhD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No